CLINICAL TRIAL: NCT02385955
Title: Prospective Multicenter Phase II Study of Myeloablative Double Unit Umbilical Cord Blood Transplantation in Adult Patients With Hematologic Malignancies
Brief Title: Phase II Study of Myeloablative Double Unit Umbilical Cord Blood Transplantation in Adult Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: The Korean Society of Blood and Marrow Transplantation (Other)
Responsible Party: Principal Investigator, Sung-Soo Yoon, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSBMT200809
Record Dates: First submitted 2015-01-20; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Myeloablative dUCBT (Experimental): Myeloablative conditioning with (1) TBI, cyclophosphamide, and cytarabine, or (2) thiotepa, busulfan, and fludarabine, followed by double unit umbilical cord blood transplant
  Interventions: Procedure: Myeloablative double unit cord blood transplantation

INTERVENTIONS:
Procedure: Myeloablative double unit cord blood transplantation — Two myeloablative conditioning regimens will be used in this study: (1) total body irradation (TBI, 12Gy), followed by cyclophosphamide (60 mg/kg/day on day -3 and -2) and cytarabine (3 g/m2 every 12 hours on day -5 and -4), or (2) thiotepa (5 mg/kg/day on day -7 and -6), busulfan (3.2 mg/kg/day on day -5, -4, and -3), and fludarabine (50 mg/m2/day on day -5, -4, and -3).

SUMMARY:
This study aimed to evaluate the efficacy and safety of myeloablative double unit umbilical cord blood transplantation (dUCBT) in adult patients with hematologic malignancies. Two myeloablative conditioning regimens will be used in this study: (1) total body irradation (TBI), cyclophosphamide, and cytarabine, or (2) thiotepa, busulfan, and fludarabine.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic malignancies requiring hematopoietic stem cell transplantation: (1) high risk acute myeloid leukemia in remission, (2) high risk acute lymphoblastic leukemia in remission, or (3) IPSS intermediate-2, high, or transfusion-dependent myelodysplastic syndrome
* Patients who have suitable cord blood units for dUCBT
* Patients with ECOG performance status 0-1
* Patients with adequate organ function: lung, kidney, liver, heart, etc.
* Informed consent

Exclusion Criteria:

* Patients who can receive hematopoietic stem cell transplantation from HLA-matched sibling or unrelated donors
* Patients who have anti-HLA antibodies
* Patients with any evidence of central nervous system (CNS) involvement of disease
* Patients with uncontrolled diabetes
* Patients with uncontrolled hypertension
* Patients with any evidence of active infection
* Positive for human immunodeficiency virus (HIV)
* Previous history of other malignancy within 5 years (Basal cell carcinoma of skin, cervical carcinoma in situ, and differentiated thyroid carcinoma with curative resection are permitted.)
* Women who are pregnant or breastfeeding
* Patients with previous history of allogeneic stem cell transplantation
* Patients with major psychotic disorder or drug/alcohol abuser
* Inappropriate patients according to the investigators' opinion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years

SECONDARY OUTCOMES:
Progression-free survival | 2 years
Time to relapse or progression | 2 years
Time to engraftment | 2 years
Acute graft-versus-host disease | 2 years
Chronic graft-versus-host disease | 2 years
Non-relapse mortality | 2 years
Other transplant-related serious adverse events | 2 years

REFERENCES:
- [Background] Takahashi S, Ooi J, Tomonari A, Konuma T, Tsukada N, Oiwa-Monna M, Fukuno K, Uchiyama M, Takasugi K, Iseki T, Tojo A, Yamaguchi T, Asano S. Comparative single-institute analysis of cord blood transplantation from unrelated donors with bone marrow or peripheral blood stem-cell transplants from related donors in adult patients with hematologic malignancies after myeloablative conditioning regimen. Blood. 2007 Feb 1;109(3):1322-30. doi: 10.1182/blood-2006-04-020172. Epub 2006 Oct 12. PMID 17038536
- [Background] Mori T, Tanaka M, Kobayashi T, Ohashi K, Fujisawa S, Yokota A, Fujita H, Nakaseko C, Sakura T, Nannya Y, Takahashi S, Kanamori H, Kanda Y, Sakamaki H, Okamoto S; Kanto Study Group for Cell Therapy. Prospective multicenter study of single-unit cord blood transplantation with myeloablative conditioning for adult patients with high-risk hematologic malignancies. Biol Blood Marrow Transplant. 2013 Mar;19(3):486-91. doi: 10.1016/j.bbmt.2012.12.007. Epub 2012 Dec 16. PMID 23253560
- [Background] Sanz J, Boluda JC, Martin C, Gonzalez M, Ferra C, Serrano D, de Heredia CD, Barrenetxea C, Martinez AM, Solano C, Sanz MA, Sanz GF; Grupo Espanol de Trasplante Hematopoyetico y Terapia Celular (GETH). Single-unit umbilical cord blood transplantation from unrelated donors in patients with hematological malignancy using busulfan, thiotepa, fludarabine and ATG as myeloablative conditioning regimen. Bone Marrow Transplant. 2012 Oct;47(10):1287-93. doi: 10.1038/bmt.2012.13. Epub 2012 Feb 13. PMID 22327127
- [Background] Ruggeri A, Sanz G, Bittencourt H, Sanz J, Rambaldi A, Volt F, Yakoub-Agha I, Ribera JM, Mannone L, Sierra J, Mohty M, Solano C, Nabhan S, Arcese W, Gluckman E, Labopin M, Rocha V; Eurocord and Acute Leukemia Working Party of European Blood and Marrow Transplant Group. Comparison of outcomes after single or double cord blood transplantation in adults with acute leukemia using different types of myeloablative conditioning regimen, a retrospective study on behalf of Eurocord and the Acute Leukemia Working Party of EBMT. Leukemia. 2014 Apr;28(4):779-86. doi: 10.1038/leu.2013.259. Epub 2013 Sep 5. PMID 24005245